CLINICAL TRIAL: NCT02546778
Title: Effects of Radiofrequency on Located Adiposity: A Pilot Study
Brief Title: Effects of Radiofrequency on Located Adiposity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Patricia Viana da Rosa, Adjunct Professor, Federal University of Health Science of Porto Alegre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23686013.9.0000.5345
Record Dates: First submitted 2015-08-27; First posted 2015-09-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Adiposity
Keywords: Radio frequency; Female; Humans; Esthetics
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dermosux RF (Experimental): The group received the radio frequency for 20 minutes with the frequency of 1 MHz with 40 W.
  Interventions: Device: Dermosux RF

INTERVENTIONS:
Device: Dermosux RF — The radio frequency was used for 20 min in the abdomen and flanks, once per week for 7 weeks.

SUMMARY:
Nowadays increasingly quest for improved physical appearance, gradually developing the medicine of beauty, where the radio fits as an additional tool in helping some aging processes and maintenance of body shape. The aim of this study was to evaluate and compare the changes in the thickness of adipose tissue and blood levels of some biochemical markers of sedentary and active women who underwent radio frequency technique via ultrasound imaging and laboratory tests. Seven (7) sessions were held, each lasting 20 minutes each, 22 volunteers allocated into two groups, sedentary and physically active. Measures ultrasound image were collected at baseline, pre-treatment and post-treatment period period and serum biochemical parameters (lipid profile, liver and kidney) for the pre-treatment and post-treatment.

DETAILED DESCRIPTION:
The demand for treatments for localized adiposity reduction increasingly gaining ground in beauty clinics due to the constant search for the perfect body and the current standards of beauty. The localized adiposity is characterized by a hypertrophy of unilocular fat cells that occurs in some parts of the body, especially the flanks and abdomen and often food programs combined with physical activity are not enough and requires a complementary treatment for redefinition of body shapes. The radio frequency is a non-invasive technique that emits electromagnetic waves generate heat in the skin layers. The technique is indicated for the treatment of edema fibro geloid (EGF), wrinkles, sagging and is also observed lipolytic effect acting directly at the level of accumulated fat cells helping to reduce the fat layer. With this vision, the investigators seek to evaluate the effects of Radio Frequency on localized f in patients who have this fat in the abdominal region, comparing a group of sedentary women with a group of women engaged in physical activities. Also will evaluate biochemical and anthropometric parameters so that they can provide indications about the effects of radio frequency in the human body.

This is a pilot study. The sample will consist of 30 females volunteers who participate, respecting the criteria for inclusion and exclusion previously cited by reading and signing the Informed Consent and Clarified.

The sample consists of 30 participants, divided into two groups, with 15 individuals will be regular exercise practitioners and 15 are sedentary, with participants from each group will undergo a 4-week control period between the first (base period) and second (pre-treatment) evaluations. Participants will be instructed to not change their respective routine activities.

For physical activity practitioner should perform at least 150 minutes of aerobic exercise of moderate intensity in the week, or at least 75 minutes of vigorous physical activity, or even that combine physical activity of moderate and vigorous intensity during the week. Both groups will make 12 sessions on individual radio frequency applications, twice a week, total of 6 weeks treatment.

To monitor the results, diagnostic ultrasound will be used to measure the fat layer. To collect the individual will be in the supine position with a pillow under the lumbar spine. The head will be positioned above the navel and the fat thickness is measured from the inner layer of the skin to the aponeurosis of the rectus abdominis muscle in the middle of the Alba line area. To measure the fatty layer of flanks the head that was in the umbilicus will be displaced laterally with the individual still in the supine position. The head is in the transverse plane will be asked to the individual who holds the air on exhalation to collect the image. The fat thickness measurements are made with a linear probe (7.5 MHz) with a depth of 4 to 5cm. The parameters used in this study have been previously tested and showed no health risk.

Among the methods used for assessing body composition, electrical bioimpedance has been widely used, especially by high speed in processing information, being a noninvasive method, practical, reproducible, which estimates, in addition to body components, the distribution of fluid in the intracellular and extracellular spaces, as well as the quality, size and cell integrity. For assessment of body composition, Bioelectrical impedance analysis (BIA) technique is based on the model of a cylindrical conductor with length and uniform and homogeneous cross-cutting area, to which the human body resembles. Evaluations shall be performed by a professional with training and experience in this type of analysis. For the examination, will be used Maltron BF-900 model unit and will be adopted the protocol recommendations proposed by the European Society for Clinical Nutrition and Metabolism:

* Assess body mass and height of the individual at the time of examination;
* Individual fasting and not drinking alcohol for at least 8 hours;
* Urinate before the exam;
* Do not perform physical exercise in the eight hours before the test;
* No injury to the skin where the electrode will be;
* Clean the skin with alcohol;
* Position the electrodes always on the same side of the body;
* Minimum of 5 cm distance between the electrodes;
* Separated from the stem by arms 30 and legs apart by 45 °;
* Environment should be neutral (no electric or magnetic field);
* Notice the shape of the body to the risk of any possible anomaly (edema, amputation, atrophy, scoliosis, dystrophy);
* In case of obesity, use of electricity insulating material (towel, for example) between the arm and torso, and between the thighs;
* When prostheses or implants, to measure the opposite side;
* Do not use metal objects in the examination as earrings, bracelets, watches and the like.

It is not indicated for individuals who have pacemaker and who are in pregnancy.

Anthropometric measurements will be measured by a previously trained evaluator. The height is determined by the balance rule coupled with a degree in 1 mm, with the individual back to this, in an upright standing position, feet together, and trying to put the posterior surface of heels, pelvic and shoulder girdle in contact with the instrument. Prior to the first session and after the last session will be measured body weight, skin suprailiac and abdominal folds, waist circumference, waist circumference, hip circumference and waist-hip ratio calculation.

Body weight will be measured through traditional mechanical scale with 100g graduation, with front man for the same, in the upright position, feet together, wearing light clothes and without shoes. Based on these two measurements will be done calculating the Body Mass Index, kg ÷ height x height.

The skinfold measure used to estimate the percentage of body fat will be taken using caliper. The supra-iliac and abdominal folds will be measured. The suprailiac preaches will be measured, taking as anatomical reference the iliac crest, in an oblique direction to the longitudinal axis of the body, plying middle region located between the last rib and the iliac crest on the medial axillary line. Since the abdominal crease is measured as taking anatomical reference umbilicus, plying up the region located 1 to 3 cm to the right of scar parallel to the longitudinal axis of the body.

The ratio of waist to hip index is the result of the equation that divides the circumference of the abdomen (cm) by hip circumference (cm). The measurement of waist circumference will be measured with the individual standing upright during the expiratory phase of respiration, using flexible measuring tape 1.5m, accurate to one decimal place, with ribbon positioned parallel to the floor, at least measured between the iliac crest and the last rib.

In Radio Frequency procedure will be used Dermosux RF equipment to decrease localized fat in the abdomen and flanks. The parameters are: maximum power of 50 Watts at a frequency of 1 MHz and will take place the measurement of skin temperature with a digital thermometer, keeping always between 40 - 42 ° C in the quadrants of the abdominal and flank region. The handle is used with continuous and repetitive movements with light pressure. A glycerin oil film over the treatment area as coupling means will be used.

The sessions will be held 2 times a week for six consecutive weeks. The time of each session will be around 40 minutes, and will be 10 minutes in the area for median-right and another 10 minutes in the area for median-left with the patient in the supine position. With the patient in the lateral decubitus will apply an additional 10 minutes on the right flank region and 10 minutes on the left flank region. The schedule of sessions will be marked in accordance with the provision of the sample. It will also be directed at the first session the importance of voluntary not change eating habits or daily lifestyle habits such as physical activity, smoking and alcohol.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary
* physically active

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Use of radio frequency reduce the layer of fat in abdominal area | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laura P Bem, Principal Investigator — Federal University of Health Science of Porto Alegre